CLINICAL TRIAL: NCT05079672
Title: Efficacy and Safety of Dexmedetomidine in the Analgesic Prophylaxis , in Patients Undergoing Cardiovascular Surgery: Randomized Clinical Trial
Brief Title: Efficacy and Safety of Dexmedetomidine in the Analgesic Prophylaxis , in Patients Undergoing Cardiovascular Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Luiz Antonio M. Cesar, Associated Professor of Cardiology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SDCDT014/19/113
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Cardiopathy; Coronary Artery Disease; Valve Heart Disease; Pain
Keywords: Dexmedetomidine; Cardiac surgery; Analgesia
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease; Heart Valve Diseases; Pain; Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group Dexmedetomidine (Active Comparator): The patient will receive Dexmedetomidine, at the rate of 0,3μg/ kg/h, in continuous intravenous infusion from the initiation of the anesthesia up to the end of the procedure, except during the cardiopulmonary by-pass.
  Interventions: Drug: Dexmedetomidine
- Group 0,9% Saline (Placebo Comparator): The patient will receive a 0,9% saline, in continuous intravenous infusion, from the initiation of the anesthesia up to the end of the procedure, except during the cardiopulmonary by-pass.
  Interventions: Drug: 0,9% Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine injectable solution, at the rate of 0,3μg/ kg/h, will be infused from the initiation of the anesthesia up to the end of the procedure, except during the cardiopulmonary by-pass.
  Arms: Group Dexmedetomidine
Drug: 0,9% Saline — Saline 0,9% will be infused from the initiation of the anesthesia up to the end of the procedure, except during the cardiopulmonary by- pass.
  Arms: Group 0,9% Saline

SUMMARY:
Acute pain is one of the complications after cardiothoracic surgeries . It can delay patients´recovery and may increase patients´morbity and mortality. This study intends to evaluate Dexmedetomidine, a highly selective α- 2 receptor agonist, that is currently applied safely and efficiently in intraoperative cardiac surgery. It has analgesic, sedative, anxiolytic and sympatholytic properties, without respiratory- depressant effect. The aim of this study is to investigate whether the intraoperative use of dexmedetomidine is better than the standard analgesia used in the intraoperative period to reduce pain and the consequences of it.

DETAILED DESCRIPTION:
This project is a prospective, double-blinded and randomized clinical trial. Eligible participants are assigned in a 1:1 ratio to either the intervention group (Group Dexmedetomidine) or control group (Group Saline 0,9%), after written informed consent to be obtained. The patients will undergo elective cardiac surgery, with extracorporeal circulation.

In the operating room, patients will be monitored for pulse oximetry, invasive blood pressure, electrocardiograms, capnography, central venous pressure and nasopharyngeal temperature probe. Induction of anesthesia is performed with intravenous midazolam, fentanyl, etomidate and neuromuscular blocking agent. Anesthesia is maintained with sevoflurane. Dexmedetomidine, at the rate of 0,3μg/ kg/h, or placebo will be infused from the initiation of the anesthesia up to the end of the procedure, except during the cardiopulmonary by-pass. Placebo is a 0,9% saline. The follow up of the assessment of the groups will extend to the postoperative ICU, where data will be collected, during the first 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old and who are undergoing cardiac procedures (coronary artery bypass, valve replacement or combined procedure), with cardiopulmonary by- pass.

Exclusion Criteria:

* Congenital heart disease
* Infective endocarditis
* Acute myocardial infarction (<two weeks)
* Pregnancy
* Cancer
* Left ventricle ejection fraction < 40%
* Cardiogenic shock
* Emergent procedure
* Use of vasopressor and/or inotrope, in the preoperative
* Liver disfunction
* Renal replacement therapy
* Nephrectomy
* Previous renal transplantation
* Patients who are participating in another clinical research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Pain 24 hours after cardiac surgery. | 24 hours after the cardiac surgery.
  The assessment of pain intensity, in patients with self- reporting, will be done by: Numeric Rating Scale (NRS) 0- 10. Possible score range from 0 (no pain) to 10 (worst pain ever ). The assessment of pain intensity, in patients on mechanical ventilation, will be done by: Behavioral Pain Scale, through facial expression (score 1-4), upper limb movement (score 1-5) and compliance with mechanical ventilation (score 1-3). Possible score range from 3 (no pain) to 12 (maximum pain).

SECONDARY OUTCOMES:
Opioid consumption. | During the first 24 hours.
  Opioid used for the pain control. This will be noted in the medical record.

OTHER OUTCOMES:
Time from the end of surgery to extubation. | During the first 24 hours.
  This interval will be observed if the patient is not extubated at the end of the surgery. This will be noted in the medical record.
Bleeding. | During the first 24 hours.
  Bleeding after the surgery. This will be noted in the medical record.
Cardiac arrhythmias. | During the first 24 hours.
  Occurrence of cardiac arrhythmias. This will be noted in the medical record.
Serum creatinine and urea. | During the first 24 hours.
  The serum level of creatinine and urea will be observed, in the usual daily measure. This will be noted in the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Antônio Machado César, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Nova Esperança University Hospital, João Pessoa, Paraíba
  - Heart Institute (InCor), Univ. of Sao Paulo Medical School, São Paulo

IPD SHARING:
Plan to Share IPD: No
This will be decided, after data collection stars.

REFERENCES:
- [Background] Kundra S, Taneja S, Choudhary AK, Katyal S, Garg I, Roy R. Effect of a low-dose dexmedetomidine infusion on intraoperative hemodynamics, anesthetic requirements and recovery profile in patients undergoing lumbar spine surgery. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):248-253. doi: 10.4103/joacp.JOACP_338_18. PMID 31303717
- [Background] Bielka K, Kuchyn I, Babych V, Martycshenko K, Inozemtsev O. Dexmedetomidine infusion as an analgesic adjuvant during laparoscopic small es, Cyrillicholecystectomy: a randomized controlled study. BMC Anesthesiol. 2018 Apr 20;18(1):44. doi: 10.1186/s12871-018-0508-6. PMID 29678158
- [Background] Talke P, Chen R, Thomas B, Aggarwall A, Gottlieb A, Thorborg P, Heard S, Cheung A, Son SL, Kallio A. The hemodynamic and adrenergic effects of perioperative dexmedetomidine infusion after vascular surgery. Anesth Analg. 2000 Apr;90(4):834-9. doi: 10.1097/00000539-200004000-00011. PMID 10735784
- [Background] Aho MS, Erkola OA, Scheinin H, Lehtinen AM, Korttila KT. Effect of intravenously administered dexmedetomidine on pain after laparoscopic tubal ligation. Anesth Analg. 1991 Aug;73(2):112-8. doi: 10.1213/00000539-199108000-00002. PMID 1854025
- [Background] Carollo DS, Nossaman BD, Ramadhyani U. Dexmedetomidine: a review of clinical applications. Curr Opin Anaesthesiol. 2008 Aug;21(4):457-61. doi: 10.1097/ACO.0b013e328305e3ef. PMID 18660652
- [Background] Kotfis K, Strzelbicka M, Zegan-Baranska M, Safranow K, Brykczynski M, Zukowski M, Ely EW; POL-BPS Study Group. Validation of the behavioral pain scale to assess pain intensity in adult, intubated postcardiac surgery patients: A cohort observational study - POL-BPS. Medicine (Baltimore). 2018 Sep;97(38):e12443. doi: 10.1097/MD.0000000000012443. PMID 30235728
- [Background] Habibi V, Kiabi FH, Sharifi H. The Effect of Dexmedetomidine on the Acute Pain After Cardiothoracic Surgeries: A Systematic Review. Braz J Cardiovasc Surg. 2018 Jul-Aug;33(4):404-417. doi: 10.21470/1678-9741-2017-0253. PMID 30184039
- [Background] Hall R. Identification of inflammatory mediators and their modulation by strategies for the management of the systemic inflammatory response during cardiac surgery. J Cardiothorac Vasc Anesth. 2013 Oct;27(5):983-1033. doi: 10.1053/j.jvca.2012.09.013. Epub 2012 Dec 29. No abstract available. PMID 23276596
- [Background] Brandao PG, Lobo FR, Ramin SL, Sakr Y, Machado MN, Lobo SM. Dexmedetomidine as an Anesthetic Adjuvant in Cardiac Surgery: a Cohort Study. Braz J Cardiovasc Surg. 2016 May-Jun;31(3):213-218. doi: 10.5935/1678-9741.20160043. PMID 27737403
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256